CLINICAL TRIAL: NCT00198237
Title: Genomic and Proteomic Analysis of Docetaxel and Capecitabine as Primary Chemotherapy for Stage II-III Breast Cancer
Brief Title: Genomic & Proteomic Analysis of Docetaxel & Capecitabine as Primary Chemo for Stage II-III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0211-27
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Capecitabine

INTERVENTIONS:
Drug: docetaxel & capecitabine

SUMMARY:
The primary objective of this study is to determine the efficacy & toxicity of combined docetaxel & capecitabine as primary chemo for subjects w/ stage II-III breast cancer.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the efficacy & toxicity of combined docetaxel & capecitabine as primary chemotherapy for subjects with stage II-III breast cancer.Subjects will be randomized into one of two groups: Docetaxel followed by four cycles of docetaxel & capecitabine vs. capecitabine followed by four cycles of docetaxel and capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the breast w/ Stage II-III disease w/ a primary tumor >/=2cm or clinically palpable axillary lymph nodes.
* Pre-treatment core or incisional bx w/ adequate tissue for histology & genomic/proteomic analysis.
* Primary tumor must be bi-dimensionally measurable by physical exam or dx breast imaging. Measurements must be obtained w/in 3 wks prior to study entry.
* Adequate organ fxn:AGC>1500; Hb>/=9.0;plts>/=100K; Crt</=2.0;Cacl Crt Clr>/=50; total bili</=ULN; LFTs<2.0 ULN
* ECOG performance status 0-1
* Neg. pregnancy test

Exclusion Criteria:

* Pts may not have had definitive primary surgery.
* Metastatic breast cancer
* Any prior chemo or hormonal therapy for breast cancer
* Prior history of malignancy w/in the previous 5 yrs.
* No active unresolved infection
* No major surgery w/in 2wks of start of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-03; Study Completion 2005-12

PRIMARY OUTCOMES:
The primary objective of this study is to determine the efficacy & toxicity of combined docetaxel & capecitabine as primary chemotherapy for subjects with stage II-III breast cancer.

SECONDARY OUTCOMES:
To evaluate genomic and proteonomic changes after initial therapy with docetaxel & capecitabine as monotherapy after combined docetaxel & capecitabine therapy.
To compare pre-treatment genomic and proteomic profiles in responders and non-responders.
To compare the results of serum-based and tissue-based proteomic analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States